CLINICAL TRIAL: NCT05570695
Title: How do Alpha Oscillations Shape the Perception of Pain? - An EEG-based Neurofeedback Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Research Foundation (Other); Studienstiftung des deutschen Volkes (Unknown)
Responsible Party: Principal Investigator, Markus Ploner, Professor of Human Pain Research, Technical University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09/2022
Record Dates: First submitted 2022-09-22; First posted 2022-10-07 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Experimental Pain in Healthy Human Subjects
Keywords: pain; neurofeedback; alpha; neural oscillations; attention; brain; registered report
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Each participant will participate in 4 experimental conditions differing with respect to the administered neurofeedback training: (1) attention right training, ARTNF; (2) attention left training, ALTNF; (3) sham attention right training, ARTsham; (4) sham attention left training, ALTsham. During neurofeedback, noxious stimuli will be applied to the dorsum of the left hand using cutaneous laser stimulation (Nd:YAP laser, Stimul 1340, DEKA M.E.L.A. srl, Calenzano, Italy; stimulation settings: 4 ms duration, 7 mm stimulus diameter, 3.5 J laser intensity) while pain ratings will be recorded.
Masking Description: Double-blinding will be enabled through the usage of sham conditions which comprise an identical sequence of events as the verum conditions and participant-specific numeric codes encoding the order of conditions. During each session, these codes will automatically (1) determine the predefined training conditions and (2) generate file names. Thus, the experimenter will be blinded during data acquisition as well as during subsequent preprocessing and analysis steps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurofeedback (Experimental): Modulation of brain activity using verum and sham neurofeedback.
  Interventions: Behavioral: attention right training, ARTNF; Behavioral: attention left training, ALTNF; Behavioral: sham attention right training, ARTsham; Behavioral: sham attention left training, ALTsham

INTERVENTIONS:
Behavioral: attention right training, ARTNF — In a first verum neurofeedback condition, participants will be instructed to focus attention on their right hand and the up-regulation of alpha oscillations in the right hemisphere relative to alpha oscillations in the left hemisphere will be incentivized through neurofeedback.
Behavioral: attention left training, ALTNF — In a second verum neurofeedback condition, participants will be instructed to focus attention on their left hand and the down-regulation of right relative to left alpha oscillations will be incentivized.
Behavioral: sham attention right training, ARTsham — During the first sham neurofeedback condition, participants will be instructed to focus attention on their right hand. However, the feedback signal will not mirror their brain activity. Instead, the feedback signal and the corresponding reward of the last matching verum condition completed by a previous participant, i.e., ARTNF for ARTsham, will be replayed (yoked feedback).
Behavioral: sham attention left training, ALTsham — During the second sham neurofeedback condition, participants will be instructed to focus attention on their left hand. However, the feedback signal will not mirror their brain activity. Instead, the feedback signal and the corresponding reward of the last matching verum condition completed by a previous participant, i.e., ALTNF for ALTsham, will be replayed (yoked feedback).

SUMMARY:
Pain is closely linked to alpha oscillations (8 -13 Hz) which are thought to represent a supra-modal, top-down mediated gating mechanism that shapes sensory processing. Consequently, alpha oscillations might also shape the cerebral processing of nociceptive input and eventually the perception of pain. To test this mechanistic hypothesis, the investigators designed a sham-controlled and double-blind electroencephalography (EEG)-based neurofeedback study. In a short-term neurofeedback training protocol, healthy participants will learn to up- and downregulate somatosensory alpha oscillations using attention. Subsequently, the investigators will investigate how this manipulation impacts experimental pain applied during neurofeedback. Using Bayesian statistics and mediation analysis, the investigators will test whether alpha oscillations mediate attention effects on pain perception. This approach promises causal insights into the role of alpha oscillations in shaping pain, and thereby extends previous correlative evidence. Beyond, it can aid the development of novel, non-invasive modulatory treatment approaches for chronic pain, which are urgently needed.

The prosed study protocol has been granted in-principle acceptance from PLOS Biology and the corresponding registration can be found at the OSF online repository [www.osf.io/qbkj2].

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years
* right-handedness (laterality quotient > 60 on the Edinburgh handedness inventory)
* good command of German
* written informed consent
* attendance at both sessions and compliance with instructions throughout the experiment

Exclusion Criteria:

* pregnancy
* neurological or psychiatric diseases (e.g., epilepsy, stroke, depression, anxiety disorders)
* severe general illnesses (e.g., tumors, diabetes)
* skin diseases (e.g., dermatitis, psoriasis or eczema)
* current or recurrent pain
* regular intake of medication (aside from contraception, thyroidal, and antiallergic medication)
* surgical procedures involving the head or spinal cord
* side-effects following previous thermal stimulation
* contact to a person with a SARS-CoV-2 infection within the last 2 weeks
* current symptoms of a cold or flu

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Alpha asymmetry index (AAI) during neurofeedback | During procedure (neurofeedback)
  During neurofeedback, brain activity will be recorded continuously and the AAI will be extracted. Subsequently, AAIs will be compared between neurofeedback conditions. Details regarding the complete analysis pipeline can be found at the OSF online repository [www.osf.io/qbkj2].
Pain ratings during neurofeedback (NRS; 1: 'no pain' to 100: 'worst tolerable pain') | During procedure (neurofeedback)
  At the end of each neurofeedback trial, participants will verbally rate the perceived intensity of a cutaneous laser stimulus. Subsequently, pain ratings will be compared between neurofeedback conditions. Details regarding the complete analysis pipeline can be found at the OSF online repository [www.osf.io/qbkj2].
Pain-related brain responses during neurofeedback | During procedure (neurofeedback)
  During neurofeedback, brain activity will be recorded continuously, and the pain-related brain responses will be extracted. Subsequently, pain-related brain responses will be compared between neurofeedback conditions. Details regarding the complete analysis pipeline can be found at the OSF online repository [www.osf.io/qbkj2].

SECONDARY OUTCOMES:
Motivation to participate in the training measured by a numerical rating scale (NRS; 1: 'very low' to 7: 'very high') | Before each session
  The motivation to participate in the training will be assessed using a self-report measure.
General self-efficacy (German version of the General Self-Efficacy Scale, GSE, minimum score: 10, maximum score: 40) | Before each session
  General self-efficacy will be assessed using the German version of the General Self-efficacy Scale.
Health-related locus of control (Multidimensional Health Locus of Control Scales, MHLC, minimum score: 3, maximum score: 15) | Before each session
  The health-related locus of control will be assessed using Multidimensional Health Locus of Control Scales.
Current positive or negative affect (Positive and Negative Affect Schedule, PNAS, minimum score: 10, maximum score: 50) | Before each session
  The current positive or negative affect will be assessed using the Positive and Negative Affect Schedule.
Perceived task demand (NRS; 1: 'very low' to 7: 'very high') | After each condition
  The perceived task demand will be assessed using a self-report measure.
Effort exerted (NRS; 1: 'very low' to 7: 'very high') | After each condition
  The effort exerted will be assessed using a self-report measure.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Ploner, Prof. Dr. med., Principal Investigator — Department of Neurology, Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Department of Neurology, Klinikum rechts der Isar, Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data sets will be made available at the OSF online repository upon publication [https://osf.io/qbkj2].
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately after publication
URL: https://osf.io/qbkj2

REFERENCES:
- [Background] Ploner M, Sorg C, Gross J. Brain Rhythms of Pain. Trends Cogn Sci. 2017 Feb;21(2):100-110. doi: 10.1016/j.tics.2016.12.001. Epub 2016 Dec 23. PMID 28025007
- [Background] Ros T, Enriquez-Geppert S, Zotev V, Young KD, Wood G, Whitfield-Gabrieli S, Wan F, Vuilleumier P, Vialatte F, Van De Ville D, Todder D, Surmeli T, Sulzer JS, Strehl U, Sterman MB, Steiner NJ, Sorger B, Soekadar SR, Sitaram R, Sherlin LH, Schonenberg M, Scharnowski F, Schabus M, Rubia K, Rosa A, Reiner M, Pineda JA, Paret C, Ossadtchi A, Nicholson AA, Nan W, Minguez J, Micoulaud-Franchi JA, Mehler DMA, Luhrs M, Lubar J, Lotte F, Linden DEJ, Lewis-Peacock JA, Lebedev MA, Lanius RA, Kubler A, Kranczioch C, Koush Y, Konicar L, Kohl SH, Kober SE, Klados MA, Jeunet C, Janssen TWP, Huster RJ, Hoedlmoser K, Hirshberg LM, Heunis S, Hendler T, Hampson M, Guggisberg AG, Guggenberger R, Gruzelier JH, Gobel RW, Gninenko N, Gharabaghi A, Frewen P, Fovet T, Fernandez T, Escolano C, Ehlis AC, Drechsler R, Christopher deCharms R, Debener S, De Ridder D, Davelaar EJ, Congedo M, Cavazza M, Breteler MHM, Brandeis D, Bodurka J, Birbaumer N, Bazanova OM, Barth B, Bamidis PD, Auer T, Arns M, Thibault RT. Consensus on the reporting and experimental design of clinical and cognitive-behavioural neurofeedback studies (CRED-nf checklist). Brain. 2020 Jun 1;143(6):1674-1685. doi: 10.1093/brain/awaa009. PMID 32176800
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Sorger B, Scharnowski F, Linden DEJ, Hampson M, Young KD. Control freaks: Towards optimal selection of control conditions for fMRI neurofeedback studies. Neuroimage. 2019 Feb 1;186:256-265. doi: 10.1016/j.neuroimage.2018.11.004. Epub 2018 Nov 10. PMID 30423429
- [Background] Klimesch W, Sauseng P, Hanslmayr S. EEG alpha oscillations: the inhibition-timing hypothesis. Brain Res Rev. 2007 Jan;53(1):63-88. doi: 10.1016/j.brainresrev.2006.06.003. Epub 2006 Aug 1. PMID 16887192
- [Background] Wallston KA, Wallston BS, DeVellis R. Development of the Multidimensional Health Locus of Control (MHLC) Scales. Health Educ Monogr. 1978 Spring;6(2):160-70. doi: 10.1177/109019817800600107. PMID 689890
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Derived] Hohn VD, Tiemann L, Bott FS, May ES, Fritzen C, Nickel MM, Gil Avila C, Ploner M. Neurofeedback and attention modulate somatosensory alpha oscillations but not pain perception. PLoS Biol. 2025 Jan 23;23(1):e3002972. doi: 10.1371/journal.pbio.3002972. eCollection 2025 Jan. PMID 39847605